CLINICAL TRIAL: NCT02773381
Title: A Trial Investigating the Effect of Oral Semaglutide Compared With Placebo on Postprandial Glucose and Triglyceride Metabolism, Energy Intake, Appetite Sensations and Gastric Emptying in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN9924-4248; 2015-003998-14 (EudraCT Number); U1111-1174-1070 (Other: WHO)
Record Dates: First submitted 2016-05-13; First posted 2016-05-16 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Semaglutide 3 mg, 7 mg, 14 mg (Experimental)
  Interventions: Drug: semaglutide
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: semaglutide — Oral administration once-daily.
  Arms: Semaglutide 3 mg, 7 mg, 14 mg
Drug: placebo — Oral administration once-daily.
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the effect of oral semaglutide compared with placebo on postprandial glucose and triglyceride metabolism, energy intake, appetite sensations and gastric emptying in subjects with Type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-75 years (both inclusive) at the time of signing informed consent
* Subjects diagnosed with type 2 diabetes mellitus for at least 90 days prior to the day of screening.
* Treated with diet and exercise and/or metformin monotherapy. The metformin dose should be unchanged in a period of 30 days prior to screening
* Body mass index (BMI) between 20.0-38 kg/m^2 (both inclusive)
* HbA1c (glycosylated haemoglobin) between 6.0-9.0 % (both inclusive)

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive methods (adequate contraceptive measures as required by local regulation or practice)
* Family or personal history of Multiple Endocrine Neoplasia Type 2 or Medullary Thyroids Carcinoma
* History of pancreatitis (acute or chronic)
* Presence of clinically significant or symptoms of gastrointestinal disorders potentially affecting absorption of drugs and/or nutrients, as judged by the investigator
* History of major surgical procedures involving the stomach potentially affecting absorption of trial product (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery)
* History or presence of any clinically relevant respiratory, metabolic (including dyslipedimia, however mild dyslipidaemia, defined as screening total cholesterol below or equal to 7.8 mmol/L and screening triglyceride below or equal to 3.42 mmol/L is accepted), renal, hepatic, gastrointestinal, endocrinological conditions (except conditions associated with diabetes mellitus)
* History or presence of malignant neoplasms within the last 5 years (except basal and squamous cell skin cancer and in-situ carcinomas)
* History or presence of cardiovascular disease including stable and unstable angina, myocardial infarction, transient ischaemic attack, stroke, cardiac decompensation, clinically significant arrhythmias and conduction disorders
* Renal impairment with estimated Glomerular Filtration Rate (eGFR) below 60 mL /min as defined by CKD-EPI using IDMS for serum creatinine measurement on the day of screening
* Impaired liver function, defined as ALT above or equal to 2.5 times upper normal limit (UNL) on the day of screening
* Smoker (defined as a subject who is smoking more than 1 cigarette or the equivalent per day). During the in-patient period, the subject must be willing to completely refrain from smoking and use of nicotine substitute products
* Known or suspected alcohol abuse within 1 year from screening (defined as regular intake of more than 21 units weekly for men and 14 units weekly for women - one unit of alcohol equals about 300 mL of beer or lager, one glass (100 mL) of wine, or 25 mL spirits)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-06-02 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

PRIMARY OUTCOMES:
Area under the serum glucose concentration-time curve | At 12 weeks of treatment

SECONDARY OUTCOMES:
Ad libitum energy intake during a lunch meal (following a standardised breakfast meal) | At 12 weeks of treatment
Mean postprandial increase in serum glucose concentration | At 12 weeks of treatment
Mean postprandial increase in TG (triglycerides) concentration | At 12 weeks of treatment
Area under the paracetamol plasma concentration-time curve | At 12 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Leeds, United Kingdom

REFERENCES:
- [Result] Gibbons C, Blundell J, Tetens Hoff S, Dahl K, Bauer R, Baekdal T. Effects of oral semaglutide on energy intake, food preference, appetite, control of eating and body weight in subjects with type 2 diabetes. Diabetes Obes Metab. 2021 Feb;23(2):581-588. doi: 10.1111/dom.14255. Epub 2020 Nov 27. PMID 33184979
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com